CLINICAL TRIAL: NCT02873013
Title: Research Concerning Background Factors at Time of Diagnosis and Initial Treatment and Treatment Progress Cancer Patients in Asia
Brief Title: Asia Study Group of Prostate Cancer (A-CaP Study)
Status: Enrolling by invitation | Type: Observational
Sponsor: Japan Study Group of Prostate Cancer (Other)
Responsible Party: Principal Investigator, Hideyuki Akaza, Professor, Japan Study Group of Prostate Cancer
Other Study IDs: A-CaP2015-2026
Record Dates: First submitted 2016-07-12; First posted 2016-08-19 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; observational study
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer: About 20,000 patients who have received a histopathological diagnosis of prostate cancer from ten countries in Asia.

SUMMARY:
This study will target patients who have received a histopathological diagnosis of prostate cancer and who are undergoing treatment in various forms, including active PSA surveillance, surgical treatment, radiotherapy, endocrine therapy, and chemotherapy. The study will survey information about the patient at time of diagnosis, clinical staging, details of initial treatment, status of disease progression, and prognosis at the end point of the study. The purpose of the study is to clarify distribution of staging, the actual status of treatment choices and treatment outcomes.

DETAILED DESCRIPTION:
The A-CaP will collect information in a linkable anonymized format from all medical institutions in Asian countries participating in the study and will engage in data analysis. J-CaP which has previous experience of engaging in a similar study in 2010 wll be a sponsor for A-CaP study, the aggregated results of which have been reported. The registration period for this study will be three years followed by 7 years of follow-up study, and research will be implemented across a wider range of Asian countries, with new institutions participating for the purposes of this study. As this study will be an observational study the acquisition of data will be relatively simple, and as the content of the study will be almost identical to the study conducted by J-CaP in 2010, a system for research implementation is already established at J-CaP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a histopathological diagnosis of prostate cancer between January 1,2016,and December 31,2018.
* Patients who, having received a diagnosis within the abovementioned period, began initial treatment for prostate cancer(including active surveillance).
* Patients who are either hospitalized as outpatients.

Exclusion Criteria:

• Patients for whom information about the time of diagnosis, including histopathological diagnosis, cannot be acquired.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patients background at time of diagnosis of prostate cancer, treatment progress and prognosis with the reason for progression and subsequent treatment methods | three years
  The following items are examined for primary outcome measure.
  1. Patient background which is represented by month and year of birth; height and weight; ethnicity and family history; medical history; and name of condition/disease for which currently receiving treatment at hospital.
  2. Information pertaining to prostate cancer which is represented by PSA value at time of prostate cancer diagnosis and Gleason score.
  3. Prognosis information which is survival or death at end point of the Study.

SECONDARY OUTCOMES:
Patient QOL measured by SF-36 during treatment by comparison with A-Cap data and data in the United States and Australia | three years
  The short form 36 (SF-36) is used for an evaluation indicator of patient QOL. SF-36 includes the following eight elements.
  1. Physical functioning
  2. Role functioning Physical
  3. Bodily pain
  4. General health
  5. Vitality
  6. Social functioning
  7. Role functioning emotional
  8. Mental health
  More detailed questions are prepared under the above each eight element, which a score is produced for a quantitative outcome of the patients QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Akaza, M.D., Ph.D., Study Director — J-CaP
Locations (1):
- The University of Tokyo, Tokyo, Meguro-ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Onozawa M, Hinotsu S, Tsukamoto T, Oya M, Ogawa O, Kitamura T, Suzuki K, Naito S, Namiki M, Nishimura K, Hirao Y, Akaza H. Recent trends in the initial therapy for newly diagnosed prostate cancer in Japan. Jpn J Clin Oncol. 2014 Oct;44(10):969-81. doi: 10.1093/jjco/hyu104. Epub 2014 Aug 6. PMID 25098707
- [Background] Cooperberg MR, Hinotsu S, Namiki M, Ito K, Broering J, Carroll PR, Akaza H. Risk assessment among prostate cancer patients receiving primary androgen deprivation therapy. J Clin Oncol. 2009 Sep 10;27(26):4306-13. doi: 10.1200/JCO.2008.21.5228. Epub 2009 Aug 10. PMID 19667269